CLINICAL TRIAL: NCT05747001
Title: Retrospective Study on the Use of CENOBAMATE as Adjunctive Treatment in a Cohort of Patients Suffering From Epilepsy With Focal Onset Seizure (FOS) and Enrolled Into the Early Access Program (EAP) in Germany, France and UK
Brief Title: This is a Retrospective Study on the Use of CENOBAMATE as Adjunctive Treatment in Patients Suffering From Epilepsy in Early Access Program in Germany, France and UK
Acronym: CENOR
Status: Completed | Type: Observational
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Hippocrates Research (Other)
Responsible Party: Sponsor
Other Study IDs: 169(A)MD21350
Record Dates: First submitted 2023-01-30; First posted 2023-02-28 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-03

CONDITIONS: Focal Onset Seizure; Epilepsy
Keywords: epilepsy; FOS; cenobamate; retrospective; Early Access Program; Europe
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Cohort of patients suffering from epilepsy with Focal Onset Seizure (FOS) and enrolled into the Early Access Program (EAP) in Germany, France and UK

SUMMARY:
Cenobamate is a newly-FDA and EMA approved drug used to treat -focal-onset seizures in adult patients.

The aim of the current study is to analyse retrospectively the overall effectiveness and tolerability of cenobamate from real-world data collected in patients who partecipated in the Early Access Program (EAP) and were treated with cenobamate as adjunctive ASM.

DETAILED DESCRIPTION:
Cenobamate is a new approved drug used to treat -focal-onset seizures in adult patients. This novel tetrazole-derived carbamate seems to act primarily by two mechanisms that are commonly associated with epilepsy: cenobamate acts as a positive allosteric modulator of the GABAA ion channels and is effective in reducing repetitive neuronal firing by inhibition of voltage-gated sodium channels, although the complete mechanism of action is currently unknown.

In clinical trials, cenobamate showed also low toxicity and adverse drug reaction profile.

In European Union (EU), cenobamate received the marketing authorisation, valid throughout the EU, in March 2021. Starting from September 2020 an EAP was initiated with cenobamate as adjunctive ASM in several EU Countries such as Germany, France, and UK.

Real-world data are of importance to understand and confirm the efficacy and safety profile of drugs outside of the clinical trial setting. The aim of the current study is to analyse the overall effectiveness and tolerability of cenobamate from real-world data in a large series of patients treated with cenobamate as adjunctive ASM.

As a consequence, a retrospective collection and analysis of the data of the patients who participated in the EAP, according to the authorization received from the local regulatory or ethic authorities, was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Data from adult patients diagnosed with epilepsy with FOS participating in the EAP with cenobamate as adjunctive treatment, according to the authorization received from the local regulatory or ethic authorities will be collected and analyzed.
* Available data will be collected after obtaining consent from patient/legal representative to the processing of personal data according to the General Data Protection Regulation (GDPR) and applicable local regulation

Exclusion Criteria:

* Patient enrolled in other clinical trial during the EAP.
* Patient aged less than 18 years old.
* Patient with specific syndrome (e.g. LGS and Dravet)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients suffering from epilepsy with FOS who have been treated with cenobamate as adjunctive Anti-seizure medication (ASM) during the EAP in Germany, France and UK.
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Responder rate (%) at 3 months from the start of maintenance | 3 months from the start of maintenance
  Percentage of responder rate (defined as a ≥50% reduction from screening/baseline in focal onset seizure frequency) after 3 months of maintenance phase.

SECONDARY OUTCOMES:
Portion of responders | 1 and 3 months after start of cenobamate therapy
  Portion of responders (defined as a ≥50% and <100% reduction from screening/baseline in focal onset seizure frequency) at 1 and 3 months after start of cenobamate therapy
Portion of responders | 3, 6 and 12 months after the completion of the titration and its relation with the dosage.
  Portion of responders (defined as a ≥50% and <100% reduction from screening/baseline in focal onset seizure frequency) at 3, 6 and 12 months after the completion of the titration and its relation with the dosage.
Portion of seizure free | 1 and 3 months after start of cenobamate therapy
  Portion of seizure free (100% reduction from screening/baseline) 1 and 3 months after start of cenobamate therapy
Portion of seizure free | 3, 6 and 12 months after the completion of the titration and its relation with the dosage.
  Portion of seizure free (100% reduction from screening/baseline)3, 6 and 12 months after the completion of the titration and its relation with the dosage.
Retention rate | 1 and 3 months after start of cenobamate therapy
  Retention rate measured as percentage of patients remaining in the study and on adjunctive therapy at: 1 and 3 months after start of cenobamate therapy
Retention rate | 3, 6 and 12 months after the completion of the titration
  Retention rate measured as percentage of patients remaining in the study and on adjunctive therapy at 3, 6 and 12 months after the completion of the titration and its relation with the dosage.
No. of Adverse Reactions (ADRs), | Through study completion, an average of 2 years
  Adverse Reactions (ADRs), including DRESS, rash/hypersensitivity occurred during the EAP.
Change in Seizures Frequency | 1 and 3 months after start of cenobamate therapy
  Change in Seizures Frequency at 1 and 3 months after start of cenobamate therapy,
Change in Seizures Frequency | 3, 6 and 12 months after the completion of the titration
  Change in Seizures Frequency at 3, 6 and 12 months after the completion of the titration
Assessment of quality of life | 1 and 3 months after start of cenobamate therapy
  The quality of life was assessed through the Questionnaire Quality of Life in Epilepsy Inventory - 31 items
Assessment of quality of life | 3, 6 and 12 months after the completion of the titration
  The quality of life was assessed through the Questionnaire Quality of Life in Epilepsy Inventory - 31 items

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Rheims, Principal Investigator — Hôpital Neurologique Pierre Wertheimer - Hospices Civils de Lyon; Rhys Thoma, Principal Investigator — The Newcastle upon Tyne Hospitals NHS Trust Victoria Road, Newcastle, NE1 4LP; Felix Rosenow, Principal Investigator — Epilepsy Center Frankfurt Rhine-Main Neurocenter Schleusenweg 2 - 16 (Haus 95) 60528 Frankfurt am Main
Locations (23):
- France (8):
  - Hôpital Pierre Wertheimer - Hopsices Civils de Lyon, Bron
  - CHRU de Lille - Hôpital Roger Salengro (LILLE), Lille
  - Centre Hospitalier Universitaire (CHU) de Marseille - Hopital de la Timone, Marseille
  - CHRU de Nancy -Hopital Central, Service de Neurologie, Nancy
  - Hôpital de la Pitié-Salpêtrière, Paris
  - CHU Rennes - Pontchaillou Hospital, Rennes
  - CHU de Rouen Hôpital Charles-NicolleService de Neurophysiologie, Rouen
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg
- Germany (12):
  - Epilepsieklinik Tabor, Bernau bei Berlin
  - Epilepsy Center Bethel hospital Mara, Bielefeld
  - Klinik und Poliklinik für Epileptologie, Universitätsklinikum Bonn, Bonn
  - Neurologische Klinik, Erlangen
  - Epilepsy Center Frankfurt Rhine-Main Neurocenter, Frankfurt am Main
  - Klinik für Neurochirurgie Uniklinik Freiburg -, Freiburg im Breisgau
  - Evangelische Krankenhaus Alsterdorf, Hamburg
  - Diakonie Kork Epilepsiezentrum, Kehl
  - Epilepsiezentrum Hessen, Klinik für Neurologie, Philipps Universität Marburg - Standort Marburg, Marburg
  - Epilepsiezentrum Kleinwachau gGmbH, Radeberg
  - Neurologie - Stroke Unit - Zentrum für Epilepsie, Reinickendorf
  - Universitätsklinikum Tubingen, Tübingen
- United Kingdom (3):
  - King's College Hospital NHS Foundation Trust, London
  - UCLH NHS Trust Epilepsy Department, London
  - The Newcastle upon Tyne Hospitals, Newcastle